CLINICAL TRIAL: NCT00851877
Title: A Phase I/II Study of Nab-paclitaxel, Cisplatin and Cetuximab With Concurrent Radiation Therapy for Local-regionally Advanced Head-and-neck Squamous Cell Carcinoma
Brief Title: Nab-Paclitaxel, Cisplatin, and Cetuximab With Concurrent Radiation Therapy for Locally Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 072010-046; SCCC-112008-019; CDR0000634258
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2018-07

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Cetuximab; Cisplatin; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Radiotherapy, Intensity-Modulated

ARMS (1):
- arm one (Experimental): Nab-Paclitaxel, Cisplatin, Cetuximab, intensity-modulated radiation therapy
  Interventions: Biological: Cetuximab; Drug: Cisplatin; Drug: Nab-Paclitaxel; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Biological: Cetuximab — Cetuximab is an epidermal growth factor receptor (EGFR) inhibitor
Drug: Cisplatin — Cisplatin is an anti-cancer chemotherapy drug
  Other Names: Platinol
Drug: Nab-Paclitaxel — paclitaxel albumin-stabilized nanoparticle formulation
  Other Names: Abraxane
Radiation: intensity-modulated radiation therapy — intensity-modulated radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Radiation therapy uses high-energy x-rays to kill tumor cells. Paclitaxel albumin-stabilized nanoparticle formulation may make tumor cells more sensitive to radiation therapy. Giving radiation therapy and paclitaxel albumin-stabilized nanoparticle formulation together with cisplatin and cetuximab may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of paclitaxel albumin-stabilized nanoparticle formulation when given together with cisplatin, cetuximab, and radiation therapy to see how well they work in treating patients with locally advanced stage III or stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of paclitaxel albumin-stabilized nanoparticle formulation when combined with cisplatin, cetuximab, and radiotherapy in patients with local-regionally advanced squamous cell carcinoma of the head and neck. (Phase I)
* To evaluate the disease-free survival of patients treated with this regimen. (Phase II)

Secondary

* To identify dose-limiting toxicities in these patients treated with this regimen. (Phase I)
* To assess the safety and tolerability of this regimen. (Phases I and II)
* To assess progression-free survival and survival of patients treated with this regimen. (Phase I)
* To assess overall survival in patients treated with this regimen. (Phase II)
* To assess response rates in patients treated with this regimen. (Phases I and II)

OUTLINE: This is a multicenter, phase I dose-escalation study of paclitaxel albumin-stabilized nanoparticle formulation followed by a phase II study.

Patients receive cetuximab IV over 120 minutes in week 1. Patients then receive cetuximab IV over 60 minutes, paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes, and cisplatin IV over 60 minutes once weekly in weeks 2-8. Patients also undergo 3D conformal or intensity-modulated radiotherapy over 30 minutes on days 1-5 in weeks 2-8.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the oropharynx, hypopharynx, or larynx

  * Diagnosis based on the primary lesion and/or lymph nodes
  * Stage III or IV disease (T2, N2-3, M0 or T3-4, any N, M0)
* No primary tumor of the oral cavity, nasopharynx, sinuses, or salivary glands
* No distant metastasis by chest x-ray, CT scan, or PET/CT scan within the past 6 weeks

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* ANC > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 9.0 g/dL (transfusion or other intervention to achieve hemoglobin > 8.0 g/dL allowed)
* Bilirubin ≤ 1.5 mg/dL
* AST, ALT, and AP ≤ 2.5 times upper limit of normal
* Serum creatinine ≤ 1.5 mg/dL
* Creatinine clearance ≥ 50 mL/min
* None of the following electrolyte abnormalities grade 3-4 by CTCAE v 3.0:

  * Calcium < 7 mg/dL or > 12.5 mg/dL
  * Glucose < 40 mg/dL or > 250 mg/dL
  * Magnesium < 0.9 mg/dL or > 3 mg/dL
  * Potassium < 3 mmol/L or > 6 mmol/L
  * Sodium < 130 mmol/L or > 155 mmol/L
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other prior invasive malignancy, except for nonmelanomatous skin cancer, unless disease-free for ≥ 3 years
* No prior allergic reaction to study drugs
* No active cardiac disease, defined as any of the following:

  * Unstable angina
  * Uncontrolled hypertension
  * Myocardial infarction within the past 6 months (unless successfully treated with coronary artery bypass graft or percutaneous transluminal coronary angioplasty)
  * Uncontrolled arrhythmia
  * Congestive heart failure
  * Three or more heart-related hospitalizations within the past year
* No severe chronic obstructive pulmonary disease requiring ≥ 3 hospitalizations within the past year
* No AIDS
* No pre-existing peripheral sensory neuropathy ≥ grade 2
* No concurrent medical illnesses that would impair patient tolerance to therapy or limit survival

PRIOR CONCURRENT THERAPY:

* No prior systemic chemotherapy for this cancer

  * Prior systemic chemotherapy for a different cancer allowed
* No prior radiotherapy to the region of this cancer that would result in overlap of radiotherapy fields
* No prior initial surgical treatment (excluding diagnostic biopsy of the primary site or nodal sampling of neck disease)
* At least 48 hours since prior and no concurrent granulocytic growth factors (e.g., filgrastim [G-CSF]) during radiotherapy
* No concurrent erythropoietic growth factors (e.g., darbepoetin, erythropoietin)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-03-01 (Actual); Primary Completion 2013-10-01 (Actual); Study Completion 2015-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hak Choy, MD, Principal Investigator — Simmons Cancer Center
Locations (2):
- United States (2):
  - Baylor Research Institute, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Nab-paclitaxel 25 mg/m^2: Cetuximab 450mg/m^2 as a loading dose in week one. Cetuximab 250 mg/m^2, Cisplatin 20mg/m^2 and nab-paclitaxel 25mg/m^2 weekly, concurrent with 70 Gy in 35 fractions continuous course intensity modulated radiotherapy during weeks 2-8.
- Phase I Nab-paclitaxel 20mg/m^2; Phase II Nab-paclitaxel 20mg/m^2: Cetuximab 450mg/m^2 as a loading dose in week one. Cetuximab 250 mg/m^2, Cisplatin 20mg/m^2 and nab-paclitaxel 20mg/m^2 weekly, concurrent with 70 Gy in 35 fractions continuous course intensity modulated radiotherapy during weeks 2-8.
Period: Phase I-1
Arm/Group | Phase I Nab-paclitaxel 25 mg/m^2 | Phase I Nab-paclitaxel 20mg/m^2 | Phase II Nab-paclitaxel 20mg/m^2
Started | 7 | 0 | 0
Completed | 6 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0
Period: Phase I-2
Arm/Group | Phase I Nab-paclitaxel 25 mg/m^2 | Phase I Nab-paclitaxel 20mg/m^2 | Phase II Nab-paclitaxel 20mg/m^2
Started | 0 | 5 | 0
Completed | 0 | 5 | 0
Not Completed | 0 | 0 | 0
Period: Phase II
Arm/Group | Phase I Nab-paclitaxel 25 mg/m^2 | Phase I Nab-paclitaxel 20mg/m^2 | Phase II Nab-paclitaxel 20mg/m^2
Started | 0 | 0 | 25
Completed | 0 | 0 | 22
Not Completed | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Nab-Paclitaxel, Cisplatin, Cetuximab and Radiation Therapy: Phase I/II Cetuximab, Cisplatin and nab-paclitaxel concurrent with intensity-modulated radiotherapy.
Arm/Group | Nab-Paclitaxel, Cisplatin, Cetuximab and Radiation Therapy
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 55.5 [45 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Phase I Maximum Tolerated Dose of Nab-Paclitaxel
Description: Seven participants were assigned nab-paclitaxel in dose of 25mg/m^2. Five participants were assigned nab-paclitaxel in dose of 20mg/m^2.
Time Frame: 90 days
Population: 12 patients enrolled in the phase I study.
Measure: Number; unit: mg/m^2
Groups:
- Phase I Nab-Paclitaxel, Cisplatin, Cetuximab and Radiotherapy: Nab-Paclitaxel, Cisplatin, Cetuximab, intensity-modulated radiation therapy
  Cetuximab: Cetuximab is an epidermal growth factor receptor (EGFR) inhibitor
  Cisplatin: Cisplatin is an anti-cancer chemotherapy drug
  Nab-Paclitaxel: paclitaxel albumin-stabilized nanoparticle formulation
  intensity-modulated radiation therapy: intensity-modulated radiation therapy
Arm/Group | Phase I Nab-Paclitaxel, Cisplatin, Cetuximab and Radiotherapy
Number analyzed (Participants) | 12
mg/m^2 | 20

2. Primary Outcome: Phase II 2-year Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
  The primary endpoint of 2-year progression-free survival was measured from the date of enrollment to the first occurrence of new metastatic lesion, objective tumor progression, or death.
Time Frame: 2 year
Population: 12 patients from Phase I also participated in Phase II of this study. 25 patients enrolled in the phase II study with 3 patients withdrew from the study prior to treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase II Nab-Paclitaxel, Cisplatin, Cetuximab and Radiotherapy: Nab-Paclitaxel, Cisplatin, Cetuximab, intensity-modulated radiation therapy
  Cetuximab: Cetuximab is an epidermal growth factor receptor (EGFR) inhibitor
  Cisplatin: Cisplatin is an anti-cancer chemotherapy drug
  Nab-Paclitaxel: paclitaxel albumin-stabilized nanoparticle formulation
  intensity-modulated radiation therapy: intensity-modulated radiation therapy
Arm/Group | Phase II Nab-Paclitaxel, Cisplatin, Cetuximab and Radiotherapy
Number analyzed (Participants) | 34
percentage of participants | 60 [42 to 78]

3. Secondary Outcome: Phase II 2-year Local Control
Description: Local control is defined as the arrest cancer growth at the site of origin. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions
Time Frame: 2 year
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II Nab-Paclitaxel, Cisplatin, Cetuximab and Radiotherapy
Number analyzed (Participants) | 34
percentage of participants | 71 [55 to 87]

4. Secondary Outcome: Phase II 2-year Overall Survival
Description: median follow-up 24 months for 34 patients
Time Frame: 2 year
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Nab-Paclitaxel, Cisplatin, Cetuximab and Radiation Therapy: Nab-Paclitaxel, Cisplatin, Cetuximab, intensity-modulated radiation therapy
  Cetuximab: Cetuximab is an epidermal growth factor receptor (EGFR) inhibitor
  Cisplatin: Cisplatin is an anti-cancer chemotherapy drug
  Nab-Paclitaxel: paclitaxel albumin-stabilized nanoparticle formulation
  intensity-modulated radiation therapy: intensity-modulated radiation therapy
Arm/Group | Nab-Paclitaxel, Cisplatin, Cetuximab and Radiation Therapy
Number analyzed (Participants) | 34
percentage of participants | 68 [50 to 86]

ADVERSE EVENTS:
Time Frame: Through study completion, and average of 2 years.
Arm/Group | Nab-Paclitaxel, Cisplatin, Cetuximab and Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 1/34
Serious Adverse Events (participants affected / at risk) | 3/34
Other Adverse Events (participants affected / at risk) | 32/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Nab-Paclitaxel, Cisplatin, Cetuximab and Radiation Therapy (N=34)
Nab-Paclitaxel toxicity (Blood and lymphatic system disorders) | 1/12 (1)
grade 4 larynx edema (General disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nab-Paclitaxel, Cisplatin, Cetuximab and Radiation Therapy (N=34)
hypothyroidism (Endocrine disorders) | 7 (7)
larynx edema (General disorders) | 15 (15)
xerostomia (General disorders) | 10 (10)
fibrosis (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes